CLINICAL TRIAL: NCT00520065
Title: Comparison of Nutritional Products for People With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK06
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2007-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- #1 (Experimental): Diabetes specific enteral product
  Interventions: Other: Diabetes specific enteral product
- #2 (Active Comparator): Standard enteral feeding
  Interventions: Other: enteral nutritional formula

INTERVENTIONS:
Other: enteral nutritional formula — Meal glucose tolerance test
  Arms: #2
Other: Diabetes specific enteral product — Meal Glucose tolerance test
  Arms: #1

SUMMARY:
Part A: To compare the glucose and insulin responses of a standard tube feeding product to that of a diabetes-specific tube feeding product in individuals with type 2 diabetes.

Part B: To compare the glucose response of a standard tube feeding product to that of a diabetes-specific tube feeding product when consumed by individuals with type 2 diabetes as a sole source of nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Type 2 diabetes
* 18 to 75 years of age
* Male or non-pregnant, non-lactating female, at least 6 weeks postpartum
* If female is of childbearing potential, is practicing birth control
* BMI greater than or equal to 18.5 kg/m2 and less than 40.0 kg/m2
* Medications, such as antihyperglycemic or thyroid medications or hormone therapy, have been maintained at a constant dosage for at least two months prior to screening visit

Exclusion Criteria:

* Uses exogenous insulin for glucose control
* Type 1 diabetes
* History of diabetic ketoacidosis
* Current infection; has received corticosteroid treatment in the last 3 months, or has had surgery or received antibiotics in the last 3 weeks
* Active malignancy
* Significant cardiovascular event less than 12 weeks prior to study entry
* End stage organ failure or is status post organ transplant
* Has an active metabolic, hepatic, or gastrointestinal disease that may interfere with nutrient absorption, distribution, metabolism, or excretion excluding diabetes
* Chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV
* Taking any herbals, dietary supplements or medications, other than antihyperglycemic medications during the past four weeks that could profoundly affect blood glucose
* Fainted or experienced other adverse reactions in response to blood collection prior to this study
* Has clotting or bleeding disorders
* Allergic or intolerant to any ingredient found in the study products
* Participant in a concomitant trial that conflicts with this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Positive area under the curve (AUC) for plasma glucose and mean glucose level | 240 minutes

SECONDARY OUTCOMES:
Adjusted peak values for plasma glucose and serum insulin concentrations and positive AUC for serum insulin concentration | 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Maki, PhD, Principal Investigator — Provident Clinical Research and Consulting, Inc.
Locations (1):
- Provident Clinical Research and Consulting, Inc., Bloomington, Indiana, United States

REFERENCES:
- [Derived] Alish CJ, Garvey WT, Maki KC, Sacks GS, Hustead DS, Hegazi RA, Mustad VA. A diabetes-specific enteral formula improves glycemic variability in patients with type 2 diabetes. Diabetes Technol Ther. 2010 Jun;12(6):419-25. doi: 10.1089/dia.2009.0185. PMID 20470226